CLINICAL TRIAL: NCT02124226
Title: Low-dose Methotrexate for Change in Global Initiative for Asthma Step 5 Medications in Chronic Severe Asthma: a Randomized Controlled Trial
Brief Title: Low-dose Methotrexate for Change in Global Initiative for Asthma Step 5 Medications in Chronic Severe Asthma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universita degli Studi di Catania (Other)
Responsible Party: Principal Investigator, Riccardo Polosa, Professor, Universita degli Studi di Catania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: METGINA-005
Record Dates: First submitted 2014-04-24; First posted 2014-04-28 (Estimated); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Low Dose Methotrexate in Severe Chronic Asthma
Keywords: Chronic severe asthma, immunomodulation, methotrexate, steroids, omalizumab
MeSH Terms: interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methotrexate (Experimental): Starting dose of 7.5 mg/week + folic acid the day after for 3 weeks as add-on therapy to their existing medication. Study treatment dosage will be increased, the maintenance dose will be 10 mg/week + folic acid the day after for 27 weeks
  Interventions: Drug: Methotrexate
- Matched placebo (Placebo Comparator): Placebo pills
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methotrexate — 7.5 mg/week + folic acid the day after
  Other Names: Several brand names
  Arms: Methotrexate
Drug: Placebo — matched placebo
  Other Names: matched placebo
  Arms: Matched placebo

SUMMARY:
Patients with chronic severe asthma (CSA) have a crippling disease and current available treatments are not satisfactory. Thus, management of CSA remains a major unmet need. Although the evidence from existing randomized controlled trials fails to support a definite role for immunomodulatory drugs in these patients due to major methodologic drawbacks, findings with low-dose methotrexate (MTX) are encouraging. However, larger and well designed clinical trials are required to establish the beneficial role of MTX in CSA and for the detection of the key characteristics of those who are going to respond to this drug.

This study will be the first multi-centre RCT investigating the role of an add-on immunological modifier as a clinically useful therapeutic strategy in patients with well-phenotyped chronic severe asthma. As such, this study does not overlap with any other research currently ongoing.

DETAILED DESCRIPTION:
Patients will be recruited from the accessible asthmatic patients lists of tertiary referral centers. All patients will meet the stringent diagnostic criteria for CSA, including the requirement for the regular use of Step 5 medications (i.e. oral prednisone and/or omalizumab). The experimental design of the proposed study will take the form of a double-blind parallel-randomized placebo-controlled trial consisting of a total of eight visits including run-in and run-out periods. Patients will be randomly allocated to receive either MTX or matched placebo once a week as add-on therapy to their existing medication after run-in. Physiological, laboratory and clinical assessments will be measured regularly throughout the study and compared with baseline assessments.

We expect that MTX will reduce Step 5 medications dosage in patients with CSA without compromising the overall disease control. Improvement in several indicators of asthma severity and control will be also investigated

ELIGIBILITY:
Inclusion Criteria:

1. patients with a diagnosis of CSA taking GINA Step 5 medications (i.e. regular OCS and/or omalizumab for a minimum of 6 months);
2. failure in weaning patients completely from Step 5 medications during run-in;
3. male and female individuals age 18 - 75 years;
4. patients must be able to provide consent;

Exclusion Criteria:

1. use of immunomodulatory therapies in the preceding 3 months;
2. recent or current history of alcoholism;
3. high liver enzyme levels (greater than 2.5 times the upper limit of the normal range);
4. serum creatinine levels greater than 2.0 mg/dL
5. acute illness within 15 days of study medication administration;
6. leucopenia (below 3.0x109/L) and/or thrombocytopenia (below 100x109/L).
7. pregnancy or planning to become pregnant;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
At least 50% reduction in total dosage of GINA step 5 medications | 80 weeks

SECONDARY OUTCOMES:
clinically significant changes in clinimetric scores | 80 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Riccardo Polosa, Full Professor, Principal Investigator — Universita di Catania

REFERENCES:
- [Derived] Polosa R, Bellinvia S, Caruso M, Emma R, Alamo A, Kowalski ML, Domingo C. Weekly low-dose methotrexate for reduction of Global Initiative for Asthma Step 5 treatment in severe refractory asthma: study protocol for a randomized controlled trial. Trials. 2014 Dec 18;15:492. doi: 10.1186/1745-6215-15-492. PMID 25523634